CLINICAL TRIAL: NCT06880562
Title: Renal and Splanchnic Sympathetic Denervation as an Alternative Therapy for Resistant Hypertension and Type 2 Diabetes (RESPLASH Study)
Brief Title: The RESPLASH Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1510
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Resistant Hypertension
Keywords: Renal Sympathetic Denervation; Splanchnic Sympathetic Denervation; Hypertension; Diabetes mellitus; Catheter-based radiofrequency ablation; Lowering blood pressure; Control of glycemic levels
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CDN of Renal arteries Arm (Placebo Comparator): Catheter-based endovascular denervation (CDN) of renal arteries only, without splanchnic nerve denervation
  Interventions: Device: Renal Denervation Only
- CND of Renal Arteries and Splanchnic Nerves Arm (Experimental): Catheter-based endovascular denervation (CDN) of renal arteries and splanchnic nerves (celiac + SMA) using radiofrequency ablation
  Interventions: Device: Splanchnic Nerve Denervation; Device: Renal Denervation Only

INTERVENTIONS:
Device: Splanchnic Nerve Denervation — Catheter-based endovascular denervation (CDN) of renal arteries and splanchnic nerves (celiac + SMA) using radiofrequency ablation
  Arms: CND of Renal Arteries and Splanchnic Nerves Arm
Device: Renal Denervation Only — Catheter-based endovascular denervation (CDN) of renal arteries only, without splanchnic nerve denervation

SUMMARY:
To assess the safety and effectiveness of renal artery denervation with subsequent splanchnic nerves denervation via catheter-based radiofrequency ablation in improving blood pressure and glycemic control in patients with resistant hypertension and type 2 diabetes.

DETAILED DESCRIPTION:
The investigators propose a multicenter, prospective, single blind, randomized controlled pilot study. Patients with treatment-resistant hypertension and diabetes mellitus type 2 will be enrolled to undergo renal artery denervation with subsequent splanchnic nerves denervation for lowering blood pressure and glycemic levels.

20 patients will be randomly selected from outpatient cardiology clinics and will be assigned (1:1) to receive an FDA approved catheter-based denervation (CDN) of the renal arteries or CDN of the renal arteries with subsequent CDN of the splanchnic nerves at the level of the celiac artery and SMA. All patients will receive non-selective renal and mesenteric artery angiography prior and post CDN. All patients will undergo office systolic and diastolic blood pressure measurements, glycemic indices (HbA1c, fasting plasma insulin, C-peptide), and other laboratory assessments (plasma norepinephrine, renin, aldosterone, angiotensin II, lipids, and liver biochemistry) at baseline and outpatient follow-up visits (months 1, 3 and 6 post procedure).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75.
* History of Type 2 Diabetes Mellitus at least 5 years prior to enrollment.
* HbA1c level ≥6.5%
* Use of at least 1 oral antidiabetic agent and no changes in the last 30 days.
* History of essential hypertension with systolic Blood pressure of 160 mmHg or more (≥150 mmHg in patient with Type 2 Diabetes Mellitus), despite compliance with three of more antihypertensive drugs.
* Stable drug regimen of at least 3 antihypertensive medications with no changes for 2 weeks before enrollment.

Exclusion Criteria:

* Estimated glomerular filtration rate of less than 30 mL/min per 1.73m2.
* Type 1 diabetes mellitus.
* History of aortic pathologies such as aneurysm or dissection confirmed by immediate preprocedural angiography that would preclude the Endovascular Denervation (EDN) procedure.
* Orthostatic hypotension.
* Acute or severe systemic infection.
* History of myocardial infarction, unstable angina, or cerebrovascular accident in the previous 3 months.
* History of previous renal artery CDN.
* Pregnancy or planned pregnancy during the study period.
* Unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in office systolic and diastolic blood pressure | Baseline, 3 months
  To assess the change in office systolic and diastolic blood pressure measurements using blood pressure cuffs at baseline to 3 months after Catheter Based Denervation (CND) at 1 month and 3 month interval.

SECONDARY OUTCOMES:
Change in HbA1C | Baseline, 3 months
  To assess the change in HbA1C from baseline to 3 months after procedure and monitor the effects of renal artery denervation with subsequent splanchnic nerves denervation.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Wiley, MD, MPH, FACC, FACP, FSCAI, Principal Investigator — Tulane University
Locations (1):
- East Jefferson General Hospital, New Orleans, Louisiana, United States